CLINICAL TRIAL: NCT05466162
Title: Effects of Soft Tissue Massage Along With Mobilization Technique on Intensity of Symptoms and Functional Status of Carpal Tunnel Syndrome - A Randomized Controlled Trial
Brief Title: Soft Tissue Massage Along With Mobilization Technique on Symptoms and Functional Status of Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hamna Syed, Hamna Syed, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HamnaS
Record Dates: First submitted 2022-04-09; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: peripheral neuropathy; compression neuropathy; entrapment neuropathy; soft tissue massage; manual therapy; massage therapy; Median neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Peripheral Nervous System Diseases; Tomaculous neuropathy; Charcot-Marie-Tooth Disease; Median Neuropathy

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial. Total 60 patients will be recruited, 30 in each group that includes There will be one interventional group and one control group. Treatment will be allocated by using a random number sheet generated by SPSS software version 21. Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The interventions assigned to individual participants will be kept hidden from the outcome assessors in the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft tissue mobilization + joint and nerve Mobilization (Experimental): Soft tissue massage therapy includes Madenci hand massage technique initiate with 30-second (sec) effleurage, followed by 60- sec friction, 30-sec petrissage, 30-sec shaking, and ends with 30-sec effleurage. It takes totally of 3 min Passive mobilizations of the wrist : radio-carpal joint in flexion and extension, maintained hand in traction. (30 oscillations, 5 sets and 30 secs interval between each step)
  Inter-carpal horizontal flexion and extension. (30 oscillations, 5 sets and 30 secs interval between each step)
  . Nerve Mobilization treatment( Slider technique) followed by Shoulder will be in depression, abduction on gleno-humeral joint and rotated externally, forearm will be in a supination, elbow flexion and wrist, elbow extension and wrist, thumb, and finger flexion Treatment sessions: 3set, 10 reps, with hold for 10 secs.
  Interventions: Other: Soft tissue mobilization; Other: Joint and nerve mobilization
- joint and nerve mobilizations (Active Comparator): Inter-carpal horizontal flexion and extension. (30 oscillations, 5 sets and 30 secs interval between each step)
  . Nerve Mobilization treatment( Slider technique) followed by Shoulder will be in depression, abduction on gleno-humeral joint and rotated externally, forearm will be in a supination, elbow flexion and wrist, elbow extension and wrist, thumb, and finger flexion Treatment sessions: 3set, 10 reps, with hold for 10 secs
  Interventions: Other: Joint and nerve mobilization

INTERVENTIONS:
Other: Soft tissue mobilization — Soft tissue massage therapy includes Madenci hand massage technique initiate with 30-second (sec) effleurage, followed by 60- sec friction, 30-sec petrissage, 30-sec shaking, and ends with 30-sec effleurage. It takes totally of 3 min Passive mobilizations of the wrist : radio-carpal joint in flexion and extension, maintained hand in traction. (30 oscillations, 5 sets and 30 secs interval between each step)
  Inter-carpal horizontal flexion and extension. (30 oscillations, 5 sets and 30 secs interval between each step)
  . Nerve Mobilization treatment( Slider technique) followed by Shoulder will be in depression, abduction on gleno-humeral joint and rotated externally, forearm will be in a supination, elbow flexion and wrist, elbow extension and wrist, thumb, and finger flexion Treatment sessions: 3set, 10 reps, with hold for 10 secs
  Other Names: Nerve mobilization( Slider technique); Joint mobilization
  Arms: Soft tissue mobilization + joint and nerve Mobilization
Other: Joint and nerve mobilization — Passive mobilizations of the wrist : radio-carpal joint in flexion and extension, maintained hand in traction. (30 oscillations, 5 sets and 30 secs interval between each step)
  Inter-carpal horizontal flexion and extension. (30 oscillations, 5 sets and 30 secs interval between each step)
  Nerve Mobilization treatment( Slider technique) followed by Shoulder will be in depression, abduction on gleno-humeral joint and rotated externally, forearm will be in a supination, elbow flexion and wrist, elbow extension and wrist, thumb, and finger flexion Treatment sessions: 3set, 10 reps, with hold for 10 secs.

SUMMARY:
The objective of this experimental study is to determine the effect of soft tissue massage along with mobilization technique on intensity of pain by visual analog scale and functional status by using Jamar hand-held dynamometer, Pinch Gauge and Boston Scale for carpal tunnel syndrome questionnaire in Carpal tunnel syndrome patients. It is being conducted on patients with Carpal tunnel syndrome at Sindh Institute of Physical Medicine and Rehabilitation, Karachi and Neurological outpatient department of Dr. Ruth K. M. Pfau, Civil Hospital Karachi among Sixty participants with mild and moderate severity of Carpal Tunnel Syndrome will be randomly allocated in two groups after initial screening by a consultant physiatrist according to CTS-6 scale. Written informed consent will be taken from each participant. Group A will be treated with soft tissue massage (Medenci hand massage technique) along with joint (radiocarpal and inter-carpal) and median nerve mobilization slider technique while group B will be treated with joint (radiocarpal and inter-carpal) and median nerve mobilization slider technique only. Participant will be evaluated by visual analog pain scale, Boston scale of carpal tunnel syndrome, dynamometer and -pinch gauge, Center for Epidemiologic Studies Depression Scale and Pain Anxiety Symptoms Scale on day 1 and last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Consultant Physiatrist will be diagnosed patients of carpal tunnel syndrome on electro diagnostic test i.e. Nerve Conduction Studies.
* Mild and moderate severity of Carpal tunnel syndrome.
* Age: 18-50 years
* Both gender patients with unilateral involvement of the hand

Exclusion Criteria:

* Exclusion Criteria:

  * In electro diagnostic test, either motor or sensory deficit in the ulnar nerve and radial nerve.
  * Other Neurological problems ( cervical myelopathy, motor neuron disease like amyotrophic lateral sclerosis
  * Neoplasm around the affected arm
  * Presence of other musculoskeletal problems of upper quadrant (for example: rheumatoid arthritis or fibromyalgia, cervical radiculopathy)
  * Any recent history of trauma of upper extremity on affected side

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity on Visual Analog Scale in centimeter after sixth week | At baseline and after completion of study at after sixth week
  Visual Analog Scale can be defined as a subjective psychometric response scale used to measure distinct behavioral or physiological phenomena based on linear numerical gradient in pain intensity measurement. The patients rate their pain intensity on 0 to 10 cm where 0 cm refers 'no pain' and 10 cm refers 'most excruciating pain'. Increase in number of cm suggests worst pain.
Change in symptoms severity and functional status on scale of Boston Carpal Tunnel Questionnaire in scores | At baseline and after completion of study at after sixth week
  It is a self-administered likert scale, containing two parts, namely the symptom severity scale and the functional status scale. It is used to assess the severity of symptoms and evaluate the difficulty in implementing the designated task. Symptom severity scale contains 11 items and the functional status scale contans 8 items. Higher the score in both scales indicating higher severity and more difficulty in performing the task.
  Scoring for Symptoms severity scale:
  Less than 11 or 11 = Asymptomatic, 12 to 22 = Mild, 23-33 = Moderate, 24-44 = Severe, 45-55 = Very Severe
  Scoring for Functional status scale:
  less than 8 or 8 = Asymptomatic, 9-16 = Mild, 17-24 = Moderate, 25-32 = Severe, 33-40 = Very Severe
  The total score of both scale is calculated as the mean of the scores for the total items of scale.
Change in hand grip strength by using Jamar dynamometer | At baseline and after completion of study at sixth week
  Hand grip strength is quantify in kilogram by using Jamar dynamometer. Measurements was taken three times of each individuals and then calculated mean of these readings.
Change in pinch strength by using Pinch Gauge | At baseline and after completion of study at sixth week
  Pinch grip strength is measured in kilogram by using Pinch Gauge. Measurements was taken three times of each individuals and then calculated mean of these readings.

OTHER OUTCOMES:
Change on Pain Anxiety Symptoms Scale-20 | At baseline and after completion of study at sixth week
  A 20 items scored on a 6-point scale from 0-5. This self-reported scale is used to assess fear of pain and consist of four elements: cognitive anxiety, escape and avoidance, fearful appraisals of pain, and physiological anxiety.
  Following scoring indicates severity of symptoms:
  mild: 0 to 34 moderate: 35-67 severe 68-100
Change on Center for Epidemiological Studies-Depression scale in scores | At baseline and after completion of study at sixth week
  A 20 items self-report scale that is used to assess depression related symptoms on the basis of frequency over the past week in primary care setting.
  Following Scoring indicate severity:
  0- 10 or less than 16 : little or no symptoms of depression 16-20 mild symptoms 22 - 25 moderate symptoms 26 -60 severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Hamna Syed, DPT, Principal Investigator — Dow University of Health Sciences; Dr. Syed Imran Ahmed, MBBS,FCPS, Study Director — Sindh Institute of Physical Medicine and Rehabilitation; Dr, Naila Naeem Shahbaz, MBBS,FCPS, Study Director — Dr. Ruth K.M. Pfau Civil Hospital, Karachi; Aftab Ahmed Mirza Baig, DPT,MSAPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huisstede BM, Hoogvliet P, Franke TP, Randsdorp MS, Koes BW. Carpal Tunnel Syndrome: Effectiveness of Physical Therapy and Electrophysical Modalities. An Updated Systematic Review of Randomized Controlled Trials. Arch Phys Med Rehabil. 2018 Aug;99(8):1623-1634.e23. doi: 10.1016/j.apmr.2017.08.482. Epub 2017 Sep 20. PMID 28942118
- [Background] Klokkari D, Mamais I. Effectiveness of surgical versus conservative treatment for carpal tunnel syndrome: A systematic review, meta-analysis and qualitative analysis. Hong Kong Physiother J. 2018 Dec;38(2):91-114. doi: 10.1142/S1013702518500087. Epub 2018 Jul 2. PMID 30930582
- [Background] Iftikhar S, Javed MA, Kasuri MN. Frequency of Metabolic Syndrome and Its Components in Patients with Carpal Tunnel Syndrome. J Coll Physicians Surg Pak. 2016 May;26(5):380-3. PMID 27225142
- [Background] Papanicolaou GD, McCabe SJ, Firrell J. The prevalence and characteristics of nerve compression symptoms in the general population. J Hand Surg Am. 2001 May;26(3):460-6. doi: 10.1053/jhsu.2001.24972. PMID 11418908
- [Background] de Krom MC, Knipschild PG, Kester AD, Thijs CT, Boekkooi PF, Spaans F. Carpal tunnel syndrome: prevalence in the general population. J Clin Epidemiol. 1992 Apr;45(4):373-6. doi: 10.1016/0895-4356(92)90038-o. PMID 1569433
- [Background] Nataraj R, Evans PJ, Seitz WH Jr, Li ZM. Effects of carpal tunnel syndrome on reach-to-pinch performance. PLoS One. 2014 Mar 14;9(3):e92063. doi: 10.1371/journal.pone.0092063. eCollection 2014. PMID 24632925
- [Background] Soon B, Vicenzino B, Schmid AB, Coppieters MW. Facilitatory and inhibitory pain mechanisms are altered in patients with carpal tunnel syndrome. PLoS One. 2017 Aug 30;12(8):e0183252. doi: 10.1371/journal.pone.0183252. eCollection 2017. PMID 28854251
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240
- [Background] Aboonq MS. Pathophysiology of carpal tunnel syndrome. Neurosciences (Riyadh). 2015 Jan;20(1):4-9. PMID 25630774
- [Background] Shin YH, Yoon JO, Kim YK, Kim JK. Psychological Status Is Associated With Symptom Severity in Patients With Carpal Tunnel Syndrome. J Hand Surg Am. 2018 May;43(5):484.e1-484.e8. doi: 10.1016/j.jhsa.2017.10.031. Epub 2018 Jan 3. PMID 29305236
- [Background] Koca I, Boyaci A, Tutoglu A, Ucar M, Kocaturk O. Assessment of the effectiveness of interferential current therapy and TENS in the management of carpal tunnel syndrome: a randomized controlled study. Rheumatol Int. 2014 Dec;34(12):1639-45. doi: 10.1007/s00296-014-3005-3. Epub 2014 Apr 12. PMID 24728028
- [Background] Eftekharsadat B, Babaei-Ghazani A, Habibzadeh A. The Efficacy of 100 and 300 mg Gabapentin in the Treatment of Carpal Tunnel Syndrome. Iran J Pharm Res. 2015 Fall;14(4):1275-80. PMID 26664397
- [Background] Geler Kulcu D, Bursali C, Aktas I, Bozkurt Alp S, Unlu Ozkan F, Akpinar P. Kinesiotaping as an alternative treatment method for carpal tunnel syndrome. Turk J Med Sci. 2016 Jun 23;46(4):1042-9. doi: 10.3906/sag-1503-4. PMID 27513402
- [Background] Chung VC, Wong SY, Kung K, Zee CY, Leung WN, Chong KC, Wong M, Wong C, Griffiths SM. Electroacupuncture and wrist splinting for carpal tunnel syndrome: a randomised trial. Hong Kong Med J. 2017 Jun;23 Suppl 2(3):28-31. No abstract available. PMID 29938668
- [Background] Khosrawi S, Emadi M, Mahmoodian AE. Effectiveness of splinting and splinting plus local steroid injection in severe carpal tunnel syndrome: A Randomized control clinical trial. Adv Biomed Res. 2016 Feb 8;5:16. doi: 10.4103/2277-9175.175902. eCollection 2016. PMID 26962518
- [Background] Lewis KJ, Coppieters MW, Ross L, Hughes I, Vicenzino B, Schmid AB. Group education, night splinting and home exercises reduce conversion to surgery for carpal tunnel syndrome: a multicentre randomised trial. J Physiother. 2020 Apr;66(2):97-104. doi: 10.1016/j.jphys.2020.03.007. Epub 2020 Apr 11. PMID 32291222
- [Background] Lindstrom-Hazel D, Kratt A, Bix L. Interrater reliability of students using hand and pinch dynamometers. Am J Occup Ther. 2009 Mar-Apr;63(2):193-7. doi: 10.5014/ajot.63.2.193. PMID 19432057
- [Background] Klimek L, Bergmann KC, Biedermann T, Bousquet J, Hellings P, Jung K, Merk H, Olze H, Schlenter W, Stock P, Ring J, Wagenmann M, Wehrmann W, Mosges R, Pfaar O. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care: Position Paper of the German Society of Allergology (AeDA) and the German Society of Allergy and Clinical Immunology (DGAKI), ENT Section, in collaboration with the working group on Clinical Immunology, Allergology and Environmental Medicine of the German Society of Otorhinolaryngology, Head and Neck Surgery (DGHNOKHC). Allergo J Int. 2017;26(1):16-24. doi: 10.1007/s40629-016-0006-7. Epub 2017 Jan 19. PMID 28217433
- [Background] Madenci E, Altindag O, Koca I, Yilmaz M, Gur A. Reliability and efficacy of the new massage technique on the treatment in the patients with carpal tunnel syndrome. Rheumatol Int. 2012 Oct;32(10):3171-9. doi: 10.1007/s00296-011-2149-7. Epub 2011 Sep 28. PMID 21953301
- [Background] Dinarvand V, Abdollahi I, Raeissadat SA, Mohseni Bandpei MA, Babaee M, Talimkhani A. The Effect of Scaphoid and Hamate Mobilization on Treatment of Patients with Carpal Tunnel Syndrome. Anesth Pain Med. 2017 Oct 23;7(5):e14621. doi: 10.5812/aapm.14621. eCollection 2017 Oct. PMID 29696114
- [Background] Wolny T, Linek P. Is manual therapy based on neurodynamic techniques effective in the treatment of carpal tunnel syndrome? A randomized controlled trial. Clin Rehabil. 2019 Mar;33(3):408-417. doi: 10.1177/0269215518805213. Epub 2018 Oct 11. PMID 30306805
- [Background] Wolny T, Linek P. Neurodynamic Techniques Versus "Sham" Therapy in the Treatment of Carpal Tunnel Syndrome: A Randomized Placebo-Controlled Trial. Arch Phys Med Rehabil. 2018 May;99(5):843-854. doi: 10.1016/j.apmr.2017.12.005. Epub 2018 Jan 4. PMID 29307812
- [Background] De-la-Llave-Rincon AI, Ortega-Santiago R, Ambite-Quesada S, Gil-Crujera A, Puentedura EJ, Valenza MC, Fernandez-de-las-Penas C. Response of pain intensity to soft tissue mobilization and neurodynamic technique: a series of 18 patients with chronic carpal tunnel syndrome. J Manipulative Physiol Ther. 2012 Jul;35(6):420-7. doi: 10.1016/j.jmpt.2012.06.002. Epub 2012 Jul 31. PMID 22858234
- [Background] Fernandez-de-Las-Penas C, Cleland J, Palacios-Cena M, Fuensalida-Novo S, Pareja JA, Alonso-Blanco C. The Effectiveness of Manual Therapy Versus Surgery on Self-reported Function, Cervical Range of Motion, and Pinch Grip Force in Carpal Tunnel Syndrome: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Mar;47(3):151-161. doi: 10.2519/jospt.2017.7090. Epub 2017 Feb 3. PMID 28158963